CLINICAL TRIAL: NCT06763016
Title: The Effect of Distant Group Counseling on Sexual Myths' and Attitudes in Young Adults: A Randomized Controlled Trial
Brief Title: Distant Group Counseling and Sexual Myths and Attitudes in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Beycan Ekitli, PhD., Ph.D., Research Assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EgeTrial5
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Sexual Risk Behavior; Sexuality
Keywords: sexual myth; sexual attitude; sexual health; counseling; telemedicine; group therapy
MeSH Terms: conditions — Sexuality | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The study is a single-blind, randomized, factorial experimental type follow-up clinical trial with a control group.
  The research design and methodology were carefully planned following the Checklist for Reporting Results of Internet E-Surveys (CHERRIES) online research guide, ensuring that the study adhered to robust research protocols. The CONSORT model was applied, including its flowchart, to enhance the transparency of the study and ensure the reproducibility of the research. The study followed a randomized controlled trial (RCT) design, and participants were randomly assigned to either the intervention or control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distant group therapy (Experimental): Distant group therapy: The intervention consisted of a six-week online group sexual counseling program. Each week, participants in the intervention group attended one 60-minute cognitive-behavioral-based tele-group session through Microsoft Teams, which was supplemented with educational content shared via Instagram.
  Interventions: Behavioral: Cognitive Behavioural Theory-based group consultation
- Control (No Intervention): Any intervention applied. Following the completion of the research, the need for psychosocial support among the control group participants was assessed, and it was found that none of them in the control group required such support.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Theory-based group consultation — The sessions focused on various topics, such as sexuality, sexual health, gender roles, and sexual violence. Participants were encouraged to engage in group discussions and complete weekly tasks, which allowed them to interact and reflect on the material presented. The intervention aimed to address and challenge prevalent sexual myths, encourage open discussions about sexuality, and foster healthier sexual attitudes through evidence-based counseling.
  The content of the digital interventions was structured on the basis of a semi-structured interactive group counseling. It was supported by sharing content on Instagram, one of the most widely used social media tools of the generation representing.
  For three days a week over six weeks, informative posts were shared, asynchronous testing and self-discovery activities were carried out, and a synchronous consultation session was held once a week. The participants were connected to the live broadcast of the research team.
  Other Names: distant consultation; group consultation; cognitive-behavioral therapy
  Arms: Distant group therapy

SUMMARY:
This study investigates the impact of distant group counseling through an online platform on sexual myths and sexual attitudes among young adults. The research design and methodology were carefully planned following the Checklist for Reporting Results of Internet E-Surveys online research guide, ensuring that the study adhered to robust research protocols. The CONSORT model was applied, including its flowchart, to enhance the transparency of the study and ensure the reproducibility of the research.

The hypotheses formulated for this randomized controlled trial are as follows:

1. There is a significant difference in the Sexual Myths Scale (SMS) pretest-posttest-follow-up scores in the intervention group.
2. There is a significant difference in the Hendrick Sexual Attitudes Scale (HSAS) pretest-posttest-follow-up scores in the intervention group.
3. There is a significant difference in the SMS pretest-posttest-follow-up scores, favoring the intervention group.
4. There is a significant difference in the HSAS pretest-posttest-follow-up scores, favoring the intervention group.

DETAILED DESCRIPTION:
Data were gathered through pretest, posttest, and follow-up assessments using established scales, including information form, the Sexual Myths Scale (SMS) and the Hendrick Sexual Attitudes Scale (HSAS).

The study followed a randomized controlled trial design, and participants were randomly assigned to either the intervention or control group. The randomization process was conducted using an online randomization tool to eliminate selection bias. Participants were randomized into the control and intervention groups based on balanced distributions of gender, pretest scores from the SMS, and the HSAS. This simple single-blind randomization process was conducted using an online randomization tool to ensure unbiased group allocation. These tools were selected for their relevance to the study's objectives and were adapted for use in an online survey format. Ethical considerations were adhered to throughout the data collection process, and participants provided informed consent before participating in the study.

The intervention consisted of a six-week online group sexual counseling program. Each week, participants in the intervention group attended one 20-minute cognitive-behavioral-based tele-group session through Microsoft Teams, which was supplemented with educational content shared via Instagram.

The intervention sessions focused on various topics, such as sexuality, sexual health, gender roles, and sexual violence. Participants were encouraged to engage in group discussions and complete weekly tasks, which allowed them to interact and reflect on the material presented. The intervention aimed to address and challenge prevalent sexual myths, encourage open discussions about sexuality, and foster healthier sexual attitudes through evidence-based counseling.

To ensure clarity and usability of the surveys, a pilot test was conducted with 10 students to gather feedback on question comprehension and the overall usability of the online platform.

Outcomes:

* Significant reduction in sexual myths in the intervention group, especially in the sexual orientation, masturbation, and sexual satisfaction subdimensions.
* Improvement in sexual attitudes in the intervention group, particularly in sexual orientation and sexual satisfaction, with the control group showing no significant changes.
* Effect size analysis demonstrated a large effect of the intervention, with 38% of the total variance explained by the combined impact of the intervention and time variables.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for participation, individuals had to meet the following criteria: be between 18-29 years of age (This period is defined as 'emerging adulthood' (Arnett, 2000), volunteer for the study, possess the necessary technological resources, and not having received any previous training on sexual health education during data collection.

Exclusion Criteria:

* Have a physical or sensory impairment that would affect the ability to use online technology (e.g., history of temporal brain damage, limb loss, hearing loss, etc.), Have a psychiatric diagnosis that would affect decision-making and orientation assessment abilities, Be receiving any professional support that could potentially influence their sexual myths and attitudes when data collection process.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Sexual Myths Scale (first evaluation with posttest) | Through intervention completion, an average of 2 month
  The scale developed by Gölbaşı et al. (2016) consists of 28 items and has 8 sub-dimensions: sexual orientation (items 1-5), gender (items 6-11), age and gender (items 12-15), sexual behavior (items 16-18), masturbation (items 19-20), sexual violence (items 21-24), sexual intercourse (items 25-26) and sexual satisfaction (items 27-28). Participants mark each item on a five-point Likert-type scale. Scale score is obtained by summing the scores given to each item in the scale. The highest score that can be obtained from the scale is 140 and the lowest score is 28. The items belonging to the sub-dimensions are summed and the score for each sub-dimension is determined. The scale does not have a cut-off point, and a high score indicates that the sexual myths are also high.
Sexual Myths Scale (second evaluation with follow up) | Through intervention completion, an average of 5 month
  The scale developed by Gölbaşı et al. (2016) consists of 28 items and has 8 sub-dimensions: sexual orientation (items 1-5), gender (items 6-11), age and gender (items 12-15), sexual behavior (items 16-18), masturbation (items 19-20), sexual violence (items 21-24), sexual intercourse (items 25-26) and sexual satisfaction (items 27-28). Participants mark each item on a five-point Likert-type scale. Scale score is obtained by summing the scores given to each item in the scale. The highest score that can be obtained from the scale is 140 and the lowest score is 28. The items belonging to the sub-dimensions are summed and the score for each sub-dimension is determined. The scale does not have a cut-off point, and a high score indicates that the sexual myths are also high.
Hendrick Sexual Attitudes Scale (first evaluation with posttest) | Through intervention completion, an average of 2 months
  The Turkish validity and reliability study of this scale, which was developed by Hendrick et al. (2006) to determine sexual attitudes, was conducted by Karaçam et al. The scale consists of four sub-dimensions and includes a total of 23 items. Each item is evaluated between 1-5 points. The questions in the birth control and sharing sub-dimension of the scale are reverse scored and the total score of the scale is not considered appropriate for evaluation. The sub-dimensions of the scale are named as affirmation (items 1-10), birth control (items 11-13), sharing (items 14-18) and instrument (items 19-23). Among these, affirmation refers to indiscriminate sexuality; birth control refers to responsible and tolerant sexuality; sharing refers to idealistic sexuality; and means refers to biological and utilitarian sexuality. High scores obtained from the affirmative and instrumental sub-dimensions of the scale indicate that the individual has an ideal, healthy and balanced sexual attitude.
Hendrick Sexual Attitudes Scale (second evaluation with follow up) | Through intervention completion, an average of 5 months
  The Turkish validity and reliability study of this scale, which was developed by Hendrick et al. (2006) to determine sexual attitudes, was conducted by Karaçam et al. The scale consists of four sub-dimensions and includes a total of 23 items. Each item is evaluated between 1-5 points. The questions in the birth control and sharing sub-dimension of the scale are reverse scored and the total score of the scale is not considered appropriate for evaluation. The sub-dimensions of the scale are named as affirmation (items 1-10), birth control (items 11-13), sharing (items 14-18) and instrument (items 19-23). Among these, affirmation refers to indiscriminate sexuality; birth control refers to responsible and tolerant sexuality; sharing refers to idealistic sexuality; and means refers to biological and utilitarian sexuality. High scores obtained from the affirmative and instrumental sub-dimensions of the scale indicate that the individual has an ideal, healthy and balanced sexual attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year after publication with no end date